CLINICAL TRIAL: NCT02178033
Title: The Impact of Split Dose of Low-volume Polyethylene Glycol on Adenoma Detection Rate: a Randomized, Investigator Blind, Controlled Trial
Brief Title: The Impact of Split Dose of Low-volume Polyethylene Glycol on Adenoma Detection Rate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Valduce Hospital (Other)
Collaborators: Istituto Clinico Humanitas (Other); Istituti Ospitalieri di Cremona (Other); Nuovo Regina Margherita Hospital (Other)
Responsible Party: Principal Investigator, Franco Radaelli, MD, Valduce Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Split dose-ADR
Record Dates: First submitted 2014-06-25; First posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Colonic Adenomas
Keywords: adenoma detection rate, screening colonoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- low-volume (2L) PEG (Other): All participants will receive low-volume (2L) PEG plus ascorbic acid solution (MOVIPREP®*, Norgine, Harefield, United Kingdom); Bowel cleansing preparation is divided into two equal doses (each MOVIPREP® sachet dissolved in one liter of water, according to manufacturer's instruction). Each dose must be followed by at least 0.5 L of clear fluid at each administration, and should be taken in a maximum time of 2 hours. In this arm, both doses are taken the day before colonoscopy, starting on the evening at about 18:00. Solution intake should be completed before 22.00 h.
  Interventions: Drug: Split dose low-volume PEG solution
- Split dose low-volume PEG solution (Active Comparator): All participants will receive low-volume (2L) PEG plus ascorbic acid solution (MOVIPREP®*, Norgine, Harefield, United Kingdom); Bowel cleansing preparation is divided into two equal doses (each MOVIPREP® sachet dissolved in one liter of water, according to manufacturer's instruction). Each dose must be followed by at least 0.5 L of clear fluid at each administration, and should be taken in a maximum time of 2 hours. In this arm, the first dose is taken on the evening before colonoscopy (at about 20:00 h), the second one is taken early in the morning on the day of the procedure, starting about 4 h before the scheduled procedure time.
  Interventions: Drug: Split dose low-volume PEG solution

INTERVENTIONS:
Drug: Split dose low-volume PEG solution — All participants will receive low-volume (2L) PEG plus ascorbic acid solution (MOVIPREP®, Norgine, Harefield, United Kingdom); in the "control arm" the whole colonoscopy preparation is administered the day before colonoscopy; in the " active comparator " arm one liter of the bowel preparation is administered on the evening before the colonoscopy and the remaining liter on the day of the procedure.
  Other Names: Low-volumePEG solution used in this study: MOVIPREP®, Norgine, Harefield, United Kingdom

SUMMARY:
An adequate level of bowel preparation is crucial for the efficacy and safety of colonoscopy. Strong evidences suggest that bowel-preparation quality shows an inverse correlation with length of the interval between the end of cleansing agent intake and the start of colonoscopy (shorter intervals are associated with better preparation levels). Accordingly, the use of a split-dose administration regimen has been demonstrated to significantly improve the quality of preparation, besides patient acceptability, as compared with standard administration the day before colonoscopy. All randomized controlled trials comparing split versus standard preparations were primarily aimed at assessing the quality of colon cleansing, by means of either validated or not-validated colon cleansing scales. The impact of a split dose regimen on objective colonoscopy performance measures such as adenoma detection rate (ADR) has never been specifically and prospectively evaluated.

The present study is aimed at evaluating whether the split-dose preparation regimen is associated with an increase of adenoma detection.

For this purpose, asymptomatic subjects aged 50-69, undergoing screening colonoscopy for positive immunologic fecal occult blood test are randomized in a 1:1 ratio to receive low-volume (2L) PEG plus ascorbic acid solution either in a split-dose (study arm) or in a full-dose regimen (control arm).

Treatments are allocated using a computer-generated, randomized code list. The treatment allocation is concealed and is accomplished at the screening visit through non-research personnel who is not involved in the study. To ensure masking, the endoscopists who perform the colonoscopies are not involved in the randomization process and in the pre-procedure data collection.

In this study the the primary outcome measure was the proportion of patients with at least one adenoma (Adenoma Detection Rate) in each harm. Data on bowel cleansing, patient compliance, tolerability and acceptability were also collected.

A sample size of at least 514 patients (257 in each arm) was calculated, by hypothesizing a relative increase of 25% in the adenoma detection rate in the split dose preparation group, assuming a 40% prevalence of one or more adenoma in FIT-positive patients undergoing screening colonoscopy (significance level 0.05, 90% power).

DETAILED DESCRIPTION:
All participants will receive the same low-volume (2L) PEG plus ascorbic acid solution (MOVIPREP®*, Norgine, Harefield, United Kingdom; each liter containing 100.0 g macrogol 3350, 7.5 g sodium sulfate,2.7 g sodium chloride, 1.0 g potassium chloride, 4.7 g ascorbic acid, 5.9 g sodium ascorbate, and lemon or orange flavoring).

Patients allocated in the "control arm" will receive the whole preparation the day before colonoscopy, whereas, patient randomly allocated to the "active treatment" will take one liter of the bowel preparation the evening before the procedure and the remaining liter the day of the procedure.

Participants will also receive a standardized low-fiber diet before the colonoscopy, avoiding fruit, legumes or vegetables for 3 days before the procedure. They will have a normal breakfast and a light lunch on the day before the procedure, but no solid food will be permitted since then. Liquid food (e.g., clear soup or yoghurt) will be permitted for the evening meal. Clear fluids can be taken at any time, until 2 hours before the procedure.

Treatments are allocated using a computer-generated, randomized code list. The treatment allocation is concealed and is accomplished at the screening visit through non-research personnel who is not involved in the study. To ensure masking, the endoscopists who perform the colonoscopies are not involved in the randomization process and in the pre-procedure data collection.

Data on patient compliance, tolerability and acceptability are collected on the morning of colonoscopy, immediately before the procedure, by a nurse questioned through a standardised questionnaire. The endoscopist is not allowed to take part in the questioning or to supervise the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic subjects aged 50-69 participating to regional screening program and undergoing outpatient colonoscopy for positive immunologic fecal occult blood test.

Exclusion criteria:

* patients undergoing colonoscopy as primary screening test
* patients undergoing colonoscopy for symptoms or post-polypectomy/ cancer surveillance
* patients with history of negative large bowel endoscopy within the previous 5 years
* patients with personal history of hereditary syndromes
* patients with history of colonic resection and inflammatory bowel disease
* patients with a history of radiation therapy to abdomen or pelvis
* patients with a history of severe cardiovascular, pulmonary, liver or renal disease
* patients with unstable psychiatric illness
* patients at risk for inhalation
* patients on ant-platelet therapy or anticoagulation at the time of endoscopy procedure, preventing polyp resection
* patient with known hypersensitivity or contraindications (i.e., patients with phenylketonuria or glucose-6-phosphate dehydrogenase deficiency) to the study product
* patients who are not able or refuse to provide informed written consent

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Adenoma Detection Rate | 1 year
  Proportion of patients with at least one adenoma

SECONDARY OUTCOMES:
Advanced Adenoma Detection Rate | 1 year
  Number of patients with at least one advanced adenoma (adenoma> or =10mm and/or villous component and/or high grade dysplasia)
Flat/depressed Adenoma Detection Rate | 1 year
  proportion of patients with at least one flat/depressed adenoma
Proximal sessile serrated lesion detection rate | 1 year
  Proportion of patients with at least one proximal sessile serrated lesion
Number of adenomas per patient | 1 year
  Number of adenomas per patient
Number of advanced adenomas per patient | 1 year
  Number of advanced adenomas per patient
Number of proximal adenomas | 1 year
  Number of adenomas located in the proximal colon (right and transverse colon)
Quality of bowel preparation | 1 year
  Quality of bowel cleansing measured by the Boston Bowel Preparation Scale

CONTACTS AND LOCATIONS:
Overall Officials: Franco Radaelli, MD, Principal Investigator — Ospedale Valduce, Gastroenterology Unit, Via Dante 10, 22100, Como, Italy.
Locations (2):
- Italy (2):
  - Ospedale VAlduce, Gastroenterology Unit, Como
  - IRCCS Istituto Clinico Humanitas; Gastroenterology Unit, Milan

REFERENCES:
- [Derived] Radaelli F, Paggi S, Hassan C, Senore C, Fasoli R, Anderloni A, Buffoli F, Savarese MF, Spinzi G, Rex DK, Repici A. Split-dose preparation for colonoscopy increases adenoma detection rate: a randomised controlled trial in an organised screening programme. Gut. 2017 Feb;66(2):270-277. doi: 10.1136/gutjnl-2015-310685. Epub 2015 Dec 9. PMID 26657900